CLINICAL TRIAL: NCT05731102
Title: Students' Health and Wellbeing Study (SHOT) 2022
Brief Title: Diagnostic Survey of Mental and Substance Use Disorders Among Norwegian College and University Students
Status: Completed | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Statistics Norway (Industry); Society of Interventional Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: PDB1841
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Mental Disorders; Substance Use Disorders; Treatment; Participation
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electronic version of the Composite International Diagnostic Interview 5th version (E-CIDI 5.0) — Observational study assessing prevalence of mental and substance use disorders among college and university students

SUMMARY:
The aims of this observational survey are to 1) collect data on the prevalence of mental and substance use disorders, and 2) investigate risk factors and consequences of mental and substance use disorder

DETAILED DESCRIPTION:
This project focuses on mental health, quality of life and alcohol and substance use in students pursuing higher education. The targeted population, all Norwegian college and university students, are in an important and vulnerable period of life transitions. The overall aim of the current project is two-fold: First, the investigators will conduct a clinical assessment of mental disorders by using the newly developed electronic version of the World Health Organization (WHO) Composite International Diagnostic Interview, fifth version (CIDI 5.0), developed for the WHO World Mental Health Surveys. CIDI 5.0 is a standardized interview assessing 30-days,12 months and lifetime prevalence for several mental and substance use disorders according to diagnostic criteria in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) and International Classification of Diseases 10th edition (ICD-10). The overall aim of this will be to obtain accurate prevalence rates of disorders, as well as to validate and compare the briefer instrument used in the Students' Health and Wellbeing Study (SHOT), including the Hopkins Symptom Checklist-25 (HSCL-25). Second, the investigators will examine risk factors based on data from the SHoT, which is one of the world's largest epidemiological studies of student health.

ELIGIBILITY:
Inclusion Criteria:

* Being a fulltime college or university student
* Norwegian citizenship
* Ages 18-35 years
* Sufficient understanding of Norwegian or English to conduct the interview

Exclusion Criteria:

* None

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sexes Eligible for Study: All
Study Population: The base study population of the current study stem from the SHoT 2022 study, a large national survey of students enrolled in higher education in Norway. The SHoT 2022 was a comprehensive survey of several domains of mental health and lifestyle factors, distributed electronically through a web-based platform. In short, SHoT 2022 was conducted between February 8 and April 19, 2022, and invited all full-time Norwegian students pursuing higher education. In all, 169,572 students fulfilled the inclusion criteria, of whom 59,544 students completed the online questionnaires, yielding a response rate of 35.1%.
  When consenting to participate in the SHOT2022, the students were also asked to indicate if they wished be invited to a follow-up study of mental disorders, of whom 26,311 consented.
Sampling Method: Probability Sample
Enrollment: 9585 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of mental and substance use disorders | January 2023 to February 2023
  Mental and substance use disorders assessed in standardised diagnostic interviews employing the Composite International Diagnostic Interview (CIDI 5.0). Diagnostic criteria after ICD-10 and DSM-5.

SECONDARY OUTCOMES:
The characteristics of nonparticipants in a psychiatric diagnostic survey | January 2023 to February 2023
  Compare characteristics of participants versus nonparticipants in the survey in terms of age, gender, mental health symptoms, alcohol use, and use of health services for mental health problems. Data will be retrieved from the SHOT 2022 study, and official administrative registries and health registries.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Institute of Public Health, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Researchers may gain access to participant data by contacting the SHOT publication committee. Approval from the Norwegian Regional Committee for Medical and Health Research Ethics is a pre-requirement. The SHOT dataset is administrated by the Norwegian Institute of Public Health.
Supporting Information: Study Protocol, ICF
Time Frame: August 2023 to September 2030.
Access Criteria: Approval from the Norwegian Regional Committee for Medical and Health Research Ethics. The data must be stored in secure servers which require log in and from which no data can be extracted and copied.

REFERENCES:
- [Result] Sivertsen B, Knudsen AKS, Kirkoen B, Skogen JC, Lagerstrom BO, Lonning KJ, Kessler RC, Reneflot A. Prevalence of mental disorders among Norwegian college and university students: a population-based cross-sectional analysis. Lancet Reg Health Eur. 2023 Sep 19;34:100732. doi: 10.1016/j.lanepe.2023.100732. eCollection 2023 Nov. PMID 37927428